CLINICAL TRIAL: NCT06425367
Title: Impact of Performing a Rapid Antibiotic Susceptibility Test (MHR-SIR) on Antibiotic Therapy Adaptation in Adult Patients with Enterobacterales Bacteremia, Controlled, Randomized Cluster and Cross-over Study
Brief Title: Impact of Performing a Rapid Antibiotic Susceptibility Test on Antibiotic Therapy Adaptation in Adult Patients with Enterobacterales Bacteremia
Acronym: MHR-Blood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 650-MHR Blood
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Bacteremia
Keywords: antibiogram; bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Intervention Model Description: cluster cross-over randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MHR SIR (Experimental): rapid antibiotic susceptibility testing by diffusion on MHR-SIR (Mueller-Hinton Rapid-SIR) medium from the blood culture bottle. Antibiotic susceptibility test results are obtained 7 hours after blood culture positivity
  Interventions: Diagnostic Test: Antibiotic susceptibility testing
- MH (Active Comparator): Standard antibiotic susceptibility testing by diffusion on MH (Mueller-Hinton ) medium from the blood culture bottle Antibiotic susceptibility test results are obtained 24 hours after blood culture positivity
  Interventions: Diagnostic Test: Antibiotic susceptibility testing

INTERVENTIONS:
Diagnostic Test: Antibiotic susceptibility testing — antibiotic susceptibility testing is performed on MHR-SIR or MH medium depending on randomization

SUMMARY:
Bacteremia is defined as the presence of bacteria in the blood. They can potentially lead to life-threatening septic shock.

Effective probabilistic antibiotic therapy must therefore be initiated immediately after blood cultures have been taken.

To diagnose bacteremia, blood culture bottles must first be incubated, which allows bacterial growth and early detection. Then, as soon as the sample is positive, an antibiogram of the incriminated bacterium is carried out by inoculation on MH (Mueller Hinton) medium. This diffusion antibiogram is the reference method and is obtained 24 hours after the vial is positive, i.e. around 48 hours after blood cultures are taken.

American recommendations agree that it is crucial to use rapid diagnostic tests to obtain the antibiogram. Antibiotic susceptibility test data can be used to broaden the spectrum of antibiotics in the event of ineffective therapy. They can also be used to reduce the spectrum of broad-spectrum antibiotics. This is part of the proper use of antibiotics and the reduction of multi-resistant bacteria (MRB) or highly resistant bacteria (HRB). Finally, it is also possible to carry out an early oral relay, thus avoiding intravenous infusions and their complications, and potentially reducing hospitalization times.

The investigators have evaluated a rapid antibiogram by diffusion on MHR-SIR (Mueller-Hinton Rapid-SIR) medium from the blood culture bottle. The investigators were able to obtain antibiogram results 7 hours after blood culture positivity, with excellent correlation compared with the standard method after 24 hours incubation on MH (Mueller-Hinton). The antibiotics tested were the same as with the standard method.

Secondly, The investigators were able to evaluate prospectively the impact of diffusion antibiotic susceptibility testing on MHR-SIR medium on early modification of antibiotic therapy in bacteremia, on 167 patients Antibiotic susceptibility test data on MHR-SIR enabled us to adapt antibiotic therapy 8 hours after blood culture positivity for 74 patients (44%). Antibiotic therapy was ineffective for 30 patients (18%) and was therefore extended. It also enabled us to reduce the spectrum of antibiotic therapy, in particular through early oral relay, for 44 patients (26%).

The aim of this multicenter trial is to validate on a large scale this strategy for obtaining rapid antibiotic susceptibility test results, with significant consequences in terms of optimizing antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* Patient hospitalized in a clinical department of each participating center
* Patient managed in the context of bacteremia (microbiological criterion = positive blood culture)
* Patient with positive blood culture for Enterobacterales
* Patient affiliated to a health insurance scheme
* Patient/relative having given free, informed and express oral consent

Exclusion Criteria:

* Patients with non-enterobacterial bacteremia
* Patient under guardianship
* Patient deprived of liberty
* Patient under court protection
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Effective Antiobiotherapy | 12 hours
  percentage of patients with Enterobacterales bacteremia for whom antibiotic therapy was effective against the incriminating bacterium within 12 hours of a positive blood culture, according to the results of the antibiogram.

SECONDARY OUTCOMES:
Time Frame | 3days
  Time between blood sampling and antibiogram results
type of Antibiotherapy spectra modification | 2 days
  After obtaining the antibiogram result, was the antibiotherapy modified (Yes or No) and if yes, was it for narrowing the antibiotic spectra (yes or no)
Time necessary to modify the spectrum of probabilistic antibiotic therapy after the antibiogram results | 2 days
  in hours
time between the start of intravenous antibiotic therapy and oral antibiotics. | 1month
  in days
length of hospital stay | 1 month
  In days,

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude NGUYEN VAN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No